CLINICAL TRIAL: NCT04358354
Title: Irinotecan Plus Oxaliplatin, 5-fluorouracil and Leucovorin as First-line Treatment for Metastatic Gastric Cancer
Brief Title: Triplet Combination of Cytotoxics as First-line Treatment for Metastatic Gastric Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jian Xiao, Asso. Professor, Sixth Affiliated Hospital, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAHMO206
Record Dates: First submitted 2020-04-11; First posted 2020-04-24 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-07

CONDITIONS: Metastatic Gastric Cancer
Keywords: irinotecan
MeSH Terms: conditions — Stomach Neoplasms | interventions — Irinotecan; Oxaliplatin; Fluorouracil

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FOLFOXiri group (Experimental): Irinotecan 150 mg/m2 iv drip d1; Oxaliplatin 85 mg/m2 iv drip d1; LV 200 mg/m2 iv drip d1; 5FU 400mg/m2 iv bolus and 2400 mg/m2 civ; The regimen will be repeated every 2 weeks until disease progression or untolerable toxicity.
  Interventions: Drug: Irinotecan; Drug: Oxaliplatin; Drug: 5-fluorouracil
- FOLFOX group (Active Comparator): Oxaliplatin: 85 mg/m2 iv drip d1; LV 200 mg/m2 iv drip d1; 5FU 400mg/m2 iv bolus and 2400 mg/m2 civ 46h; The regimen will be repeated every 2 weeks until disease progression or untolerable toxicity.
  Interventions: Drug: Oxaliplatin; Drug: 5-fluorouracil

INTERVENTIONS:
Drug: Irinotecan — Irinotecan 150 mg/m2
  Other Names: CPT-11
  Arms: FOLFOXiri group
Drug: Oxaliplatin — Oxaliplatin 85 mg/m2
  Other Names: LOHP
Drug: 5-fluorouracil — 5-fluorouracil 400 mg/m2 iv bolus and 2400 mg/m2 civ 46 hours
  Other Names: 5-FU

SUMMARY:
This parallel, randomized, open-label study will evaluate the effect on overall survival of irinotecan on oxaliplatin and 5-fluorouracil (5-FU) in patients with HER2-negative and pMMR metastatic gastric cancer. Irinotecan will be administered as intravenous infusion of 150 mg/m2 every 2 weeks. Oxaliplatin will be given 85 mg/m2 and 5-FU will be given 400mg/m2 iv and 2400mg/m2 civ 48 hours fortnightly. Treatment will continue until disease progress or untolerable toxicity appears. The target sample size is 350-400 patients.

DETAILED DESCRIPTION:
Eligible patients will be randomly assigned to FOLFOXiri group and FOLFOX group. Stratification factors include ECOG PS, disease extent and pathological subtypes. Efficacy will be evaluated every 3-4 cycles with RECIST. Toxicity will be assessed with WHO CTC 3.0 every 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years old, gender is not limited;
2. Inoperable locally advanced, recurrent, and/or metastatic cancer of the stomach or gastro-esophageal junction;
3. Pathologically confirmed adenocarcinoma;
4. Expected survival time ≥ 3 months;
5. ECOG PS 0-3;
6. Adequate bone marrow function reserve: white blood cell count ≥ 3.0 × 10*9 / L, neutrophil count ≥ 1.5 × 10*9/ L; platelet count ≥ 100 ×10*9/ L; hemoglobin ≥ 90 g / L;
7. AST and ALT ≤ 2.5 times the upper limit of normal value, total bilirubin ≤ 2 times the upper limit of normal value; serum creatinine ≤ 1.5 times the upper limit of normal value;
8. Be able to understand the research process, volunteer to participate in the study, and sign an informed consent form.

Exclusion Criteria:

1. Patients known to be allergic to active or other components of chemotherapeutic drugs;
2. Patients with severe peritoneal dissemination and GI obstruction;
3. Her-2 overexprssion or d-MMR;
4. Severe or uncontrolled infections that may affect the evaluation of the study treatment or study results;
5. History of other malignant tumors in the past 5 years (except for cured cervical carcinoma in situ or basal cell carcinoma of the skin);
6. Participated in other clinical trials within 4 weeks prior to the start of the study;
7. Pregnant or lactating women, or women of childbearing age who refuse to take effective contraception during the study period.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 388 (Estimated)
Dates: Start 2020-10-22 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | 2 years
  OS is defined as the time from the date of randomization to the date of death due to any cause. Participants were censored at the last date of tumor measurement, the last date in the study drug log or the date of last follow-up.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | 1 year
  PFS is defined as the time from the date of randomization to the date of the first documentation of progressive disease or date of death, whichever occurs first. For target lesions (TL), PD was defined as at least a 20 percent (%) increase in the sum of the longest diameter (SLD) of TLs, taking as a reference the smallest SLD recorded since the treatment started, or the appearance of one or more lesions. For non-target lesions (NTL), PD was defined as an unequivocal progression of existing NTLs. Participants were censored at the last date of tumor measurement, the last date in the study drug log, or the date of last follow-up.
Percentage of Participants With Confirmed Complete Response (CR) or Partial Response (PR) Determined by Response Evaluation Criteria in Solid Tumors (RECIST) | 24 weeks
  For TLs, a CR was defined as the disappearance of all TLs and a PR was defined as at least a 30% decrease in the SLD of the TLs, taking as a reference the baseline SLD. For NTLs, a CR was defined as the disappearance of all NTLs and normalization of tumor marker levels.
Duration of Response | 1 year
  Duration of response was defined for responders as the time from the date on which the CR or PR was first recorded to the date on which PD is first noted. Participants were censored on the date of death, the date of last tumor measurement, the last date in study drug log, or the date of last follow-up.
European Organisation For the Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Core 30 (QLQ C-30) Questionnaire Scores | 2 years
  EORTC QLQ-C30: included functional scales (physical, role, cognitive, emotional, and social), global health status, symptom scales (fatigue, pain, nausea/vomiting) and single items (dyspnoea, appetite loss, insomnia, constipation/diarrhea and financial difficulties). Most questions used 4 point scale (1 'Not at all' to 4 'Very much'; 2 questions used 7-point scale (1 'very poor' to 7 'Excellent'). Scores averaged, transformed to 0-100 scale; higher score equals (=) better level of functioning or greater degree of symptoms.
EORTC Quality of Life Questionnaire-Stomach Cancer Specific (QLQ STO22) Questionnaire Scores | 2 years
  The QLQ-STO22 is a gastric cancer quality of life questionnaire. There are 22 questions concerning disease, treatment related symptoms, side effects, dysphagia, nutritional aspects, and questions about the emotional problems of gastric cancer (dysphagia, pain, reflux, eating restrictions, anxiety, dry mouth, body image, and hair loss). The questions are grouped into five scales and 4 single items which are related to the symptoms of the disease. Most questions used 4-point scale (1 'Not at all' to 4 'Very much'; 1 question was a yes or no answer). A linear transformation was used to standardize all scores and single-items to a scale of 0 to 100; higher score=better level of functioning or greater degree of symptoms.
Treatment associated toxicities | 2 years
  WHO CTC 3.0

CONTACTS AND LOCATIONS:
Overall Officials: Jian Xiao, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- The Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China